CLINICAL TRIAL: NCT04726748
Title: Economic Evaluation of Prostatic Urethral Lift (Urolift)
Brief Title: Economic Evaluation of Prostatic Urethral Lift
Acronym: ECOLIFT
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Bordeaux PharmacoEpi (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2019/12
Record Dates: First submitted 2021-01-19; First posted 2021-01-27 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Urolift cohort: 80 patients with prostatic urethral lift surgery will be included
  Interventions: Procedure: Comparisons between the Prostatic urethral lift (PUL) and the TURP/Laser cohorts; Procedure: Comparison between the Prostatic urethral lift (PUL) and the SNDS cohorts
- Transurethral Resection of the Prostate/laser cohort: 80 patients with a transurethral resection of the prostate or laser surgery (enucleation or vaporisation) will be included.
  Interventions: Procedure: Comparisons between the Prostatic urethral lift (PUL) and the TURP/Laser cohorts
- National healthcare insurance system database (SNDS) cohort: 1200 patients with any transurethral surgery (TURP/laser) will be included and randomly matched to patients of the Urolift cohort with ratio 5:1.
  Interventions: Procedure: Comparison between the Prostatic urethral lift (PUL) and the SNDS cohorts

INTERVENTIONS:
Procedure: Comparisons between the Prostatic urethral lift (PUL) and the TURP/Laser cohorts — Comparison between the PUL and the TURP/Laser cohorts will be performed after 1 year and 3 years of follow-up in a intention-to-treat analysis using:
  * a linear regression model when it involves quantitative variables,
  * a logistic regression model adjusted on potential confounding when it involves qualitative variables.
  Groups: Transurethral Resection of the Prostate/laser cohort; Urolift cohort
Procedure: Comparison between the Prostatic urethral lift (PUL) and the SNDS cohorts — Comparison between the PUL and the SNDS cohorts will be performed after 1 year and 3 years of follow-up in a intention-to-treat analysis using:
  * a linear regression model when it involves quantitative variables,
  * a logistic regression model adjusted on potential confounding when it involves qualitative variables.
  Groups: National healthcare insurance system database (SNDS) cohort; Urolift cohort

SUMMARY:
Prostatic urethral lift (Urolift) has been developed as a minimally invasive alternative to transurethral resection of the prostate with no need of general anaesthesia, less need of urinary catheter and less exposure to post-operative complication. Its efficacy and safety have been assessed by 2 clinical randomized trials with evidence of urinary symptom improvement remaining inferior to TURP but durable for 5 years. Urolift preserved overall quality of life better than TURP. Urolift has been recommended by the European Association of Urology guidelines and recognized by French authorities but cannot be financed by the hospital itself. Reimbursement of the implants by healthcare system is therefore needed for the distribution of Urolift in France.

The additional cost of the implants could be compensated by a reduced length of hospital stay and a lower rate of post-operative complications inducing healthcare expenditures. This study aims to assess if Urolift could be a cost-effective therapeutic strategy compared to transurethral surgery with 2 phases design: a field study comparing patients treated with Urolift to those treated with TURP/laser during 1 year follow-up, and an additional study comparing healthcare consumptions during 3 years follow-up between each group using data of the French National Claims Database (SNDS database).

DETAILED DESCRIPTION:
Transurethral surgery such as transurethral resection of the prostate (TURP), laser enucleation or laser vaporisation, is the first line surgical treatment for bladder outlet obstruction secondary to benign prostatic hyperplasia. Even if bipolar and laser surgery have improved surgical outcomes in terms of length of hospital stay and post-operative complications, these procedures remain associated with a significant amount of infectious and bleeding complications, as well as with some persistent side effects such as sexual dysfunction and urinary incontinence.

Prostatic urethral lift (Urolift) has been developed as a minimally invasive alternative to TURP with no need of general anaesthesia, less need of urinary catheter and less exposure to post-operative complication. Its efficacy and safety have been assessed by 2 clinical randomized trials with evidence of urinary symptom improvement remaining inferior to TURP but durable for 5 years. Urolift preserved overall quality of life better than TURP. Urolift has been recommended by the European Association of Urology guidelines and recognized by French authorities but cannot be financed by the hospital itself. Reimbursement of the implants by healthcare system is therefore needed for the distribution of Urolift in France.

The additional cost of the implants could be compensated by a reduced length of hospital stay and a lower rate of post-operative complications inducing healthcare expenditures. This study aims to assess if Urolift could be a cost-effective therapeutic strategy compared to transurethral surgery with 2 phases design: a field study comparing patients treated with Urolift to those treated with TURP/laser during 1 year follow-up, and an additional study comparing healthcare consumptions during 3 years follow-up between each group using data of the French National Claims Database (SNDS database).

ELIGIBILITY:
● The PUL and TURP/LASER cohorts:

Inclusion criteria:

* male patient aged over 50 years
* patient who experienced a PUL or TURP/Laser surgery in first line of treatment for a symptomatic BPH, with an International Prostatic Symptom Score > 13, a Peak urine flow rate < 12ml/sec on a voided volume >150ml a Prostate volume >30cc to <80 cc per ultrasound.
* patient affiliated to a French health insurance system

Exclusion criteria:

* Patient with current urinary retention, post void residual urine > 250ml,
* Patient with active urinary tract infection at time of treatment,
* Patient with previous Benign Prostatic Hyperplasia procedure,
* Patient with urethral conditions that may prevent insertion and delivery of device system into bladder,
* Patient with previous pelvic surgery or irradiation,
* Patient with history of neurogenic or atonic bladder,
* Patient with biopsy of the prostate within the past 6 weeks,
* Patient with life expectancy estimated to be less than 1 year,
* Patient with history of prostate or bladder cancer,
* Patient with PSA>10ng/ml unless prostate biopsy is negative,
* Patient under guardianship or curatorship,
* Patient intending to move abroad within 1 year after inclusion will not be included either,
* Patient participating to another interventional study on benign prostatic hyperplasia during the study.

  * The SNDS cohort:

Inclusion criteria:

* male patient affiliated to a French health insurance system
* patient aged over 50 years
* patient who experienced a TURP/Laser surgery in first line of treatment for a symptomatic BPH in the same period as patients of the PUL and TURP/LASER cohorts.

Exclusion criteria:

* Patients hospitalized in one of the 6 investigational centers and patients with a previous BPH procedure,
* patient with a previous pelvic surgery or irradiation,
* patient with history of prostate or bladder cancer within the 2 previous years,
* patient with a biopsy of the prostate within the past 6 weeks,
* patient with a short life expectancy will not be included in the cohort.

Min Age: 50 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Patients of the PUL and TURP/LASER cohorts will be identified in the SNDS through their NIR national identifier (if possible) or using a probabilistic linkage with age, hospital identifier (FINESS), date of hospitalization for the procedure and International Classification of Diseases-10 discharge diagnosis. Only patients with a 2-year history before the procedure and a 3-year follow-up after the procedure will be analysed.
Sampling Method: Non-Probability Sample
Enrollment: 1360 (Estimated)
Dates: Start 2021-04-08 (Actual); Primary Completion 2023-12-09 (Actual); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
Incremental cost per avoided complication | 4 months after the date of surgical procedure
  Incremental cost per avoided complication (based on Clavien Dindo classification) of Prostatic Urethral Lift compared with classic transurethral surgery (TURP/laser) 4 months after the surgical procedure.

SECONDARY OUTCOMES:
Incremental cost per Quality adjusted life year | 12 months after the date of surgical procedure
  The incremental cost per Quality adjusted life year of Prostatic Urethral Lift compared with classic transurethral surgery at 12 months.
Overall and specific urogenital healthcare consumptions | during 3 years after surgical procedure date
  Description of the overall and specific urogenital healthcare consumptions during the 3 years of follow-up.
  Means will be compared between two independent groups using Student's t-test when normal distribution is followed (or Mann-Whitney's test when normal distribution is not followed)
Benign prostatic hyperplasia retreatment | 12 months after surgical procedure date ; 36 months after surgical porcedure date
  Any dispensing of the following medications at 1 and 3 years after surgical procedure: alpha-blockers or 5-alpha-reductase inhibitors.
Urinary incontinence evolution | Inclusion date (date of the surgical procedure completion) ; 4 months after surgical procedure
  Urinary incontinence evolution between inclusion and 4 months after surgical procedure (Incontinence Severity Index (ISI)).
Sexual quality of life evolution | Inclusion date (date of the surgical procedure completion) ; 4 months, 12 months after surgical procedure
  Sexual quality of life evolution between inclusion, 4 months and 12 months after surgical procedure (IIEF5, Male Sexual Health Questionnaire for Ejaculatory Dysfunction (MSHQ-EjD).

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Hôpital Claude Huriez, Lille
  - CHU de Montpellier, Montpellier
  - Hôpital Cochin, Paris
  - Hôpital Lyon Sud HCL, Pierre-Bénite
  - Centre Hospitalier Universitaire de Bordeaux, Talence
  - CHRU Hopitaux de Tours, Tours

IPD SHARING:
Plan to Share IPD: No